CLINICAL TRIAL: NCT01870765
Title: Prospective Randomised Study on the Safety of Non-invasive Ventilation Versus High-flow Oxygen in Patients With Hypoxemic Respiratory Failure Undergoing Fiberoptic Bronchoscopy.
Brief Title: Safety Study of Non-invasive Ventilation Versus High-flow Oxygen in Patients With Hypoxemic Respiratory Failure Undergoing Fiberoptic Bronchoscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Stefan Kluge, PD Dr. Stefan Kluge, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV-4442
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

ARMS (2):
- non-invasive ventilation (Active Comparator): Performance of bronchoscopy during non-invasive ventilation.
  Interventions: Device: non-invasive ventilation; Procedure: fiberoptic bronchoscopy
- high-flow oxygen (Experimental): Performance of bronchoscopy during high-flow oxygen therapy.
  Interventions: Device: high-flow oxygen; Procedure: fiberoptic bronchoscopy

INTERVENTIONS:
Device: non-invasive ventilation — non-invasive ventilation via face mask
  Arms: non-invasive ventilation
Device: high-flow oxygen — high-flow oxygen via nasal cannula
  Arms: high-flow oxygen
Procedure: fiberoptic bronchoscopy — fiberoptic bronchoscopy including broncho-alveolar lavage

SUMMARY:
Bronchoscopy with broncho-alveolar lavage is a diagnostic tool in patients with pneumonia. Especially patients with acute or chronic pulmonary diseases are at risk of respiratory failure during or after bronchoscopy. It is known that in these cases bronchoscopy can be performed safely using non-invasive ventilation. It seems probable that high-flow oxygen, which is used in the treatment of patients with hypoxemic respiratory failure, is equally effective in preventing the development of respiratory failure during fiberoptic bronchoscopy while improving patient comfort. In this prospective randomised study the safety of high-flow oxygen is compared with non-invasive ventilation in patients with hypoxemic respiratory failure undergoing fiberoptic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in an intensive care unit
* indication for bronchoscopy and broncho-alveolar lavage
* presence of hypoxemic (SaO2/fraction of inspired oxygen(FiO2): 300 or less) and/or hypercapnic respiratory failure

Exclusion Criteria:

* patients already on invasive ventilation
* indication for intubation
* blocked nasopharynx
* contraindications for non-invasive ventilation or high-flow oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Mean decrease in the saturation of oxygen (SpO2) during bronchoscopy. | during fiberoptic bronchoscopy

SECONDARY OUTCOMES:
Changes in blood gases after the completion of fiberoptic bronchoscopy. | 1 hour after the completion of bronchoscopy

OTHER OUTCOMES:
Requirement of intubation after the completion of bronchoscopy. | 8 hours after the completion of bronchoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Department of Intensive Care Medicine, Hamburg, Germany

REFERENCES:
- [Result] Simon M, Braune S, Frings D, Wiontzek AK, Klose H, Kluge S. High-flow nasal cannula oxygen versus non-invasive ventilation in patients with acute hypoxaemic respiratory failure undergoing flexible bronchoscopy--a prospective randomised trial. Crit Care. 2014 Dec 22;18(6):712. doi: 10.1186/s13054-014-0712-9. PMID 25529351